CLINICAL TRIAL: NCT00100165
Title: Phase 2 Trial of the Nicotinic Agonist 3-(2,4 Dimethoxybenzylidene Anabaseine) in Schizophrenia
Brief Title: Phase 2 Trial of a Nicotinic Agonist in Schizophrenia
Acronym: DMXB-A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-0837; VISN 19 MIRECC (Other Grant/Funding Number: VA)
Record Dates: First submitted 2004-12-23; First posted 2004-12-24 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3-(2,4 dimethoxybenzylidene anabaseine) 150 mg (Experimental): Patient receives 3-(2,4 dimethoxybenzylidene anabaseine) 150 mg twice per day in a blinded capsule.
  Interventions: Drug: 3-(2,4 dimethoxybenzylidene anabaseine) 150 mg
- 3-(2,4 dimethoxybenzylidene anabaseine)75 mg (Experimental): Patient receives 3-(2,4 dimethoxybenzylidene anabaseine) 75 mg twice per day in a blinded capsule.
  Interventions: Drug: 3-(2,4 dimethoxybenzylidene anabaseine) 75 mg
- placebo (Placebo Comparator): Patient receives placebo twice per day in a blinded capsule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo by mouth twice a day for 4 weeks
  Other Names: inactive substance
  Arms: placebo
Drug: 3-(2,4 dimethoxybenzylidene anabaseine) 150 mg — 3-(2,4 dimethoxybenzylidene) 150 mg by mouth twice a day for 4 weeks
  Other Names: GTS-21
  Arms: 3-(2,4 dimethoxybenzylidene anabaseine) 150 mg
Drug: 3-(2,4 dimethoxybenzylidene anabaseine) 75 mg — 3-(2,4 dimethoxybenzylidene) 75 mg by mouth twice a day for 4 weeks
  Other Names: GTS-21
  Arms: 3-(2,4 dimethoxybenzylidene anabaseine)75 mg

SUMMARY:
The study hypothesis is that 3-2,4 dimethoxybenzylidene anabaseine (DMXB-A), an orally administered nicotinic cholinergic agonist, will improve attention and other neuropsychological dysfunctions in schizophrenia, leading to improved psychosocial outcome.

DETAILED DESCRIPTION:
The objective of the trial is to determine if dosing 3-(2,4 dimethoxybenzylidene anabaseine) twice daily for 4 weeks will improve cognition and be safe. Secondary goals are to determine if these neurocognitive effects also have effects on neurobiological paradigms previously shown to be responsive to nicotinic receptor stimulation: suppression of P50 auditory evoked response, saccadic intrusions during smooth pursuit eye movements, and hemodynamic activity in the hippocampus during smooth pursuit eye movements as measured by functional magnetic resonance imaging. The purpose of these neurobiological measures is to assess whether the response to 3-(2,4 dimethoxybenzylidene anabaseine) is consistent with activation of nicotinic receptors. In addition, the investigators will assess clinical response using a battery of clinical assessment scales and assessments of daily living functions. The purpose of these assessments is to address the FDA requirement of a clinical effect beyond change in laboratory neuropsychological performance. This study and the subsequent two studies will also include assessments of the safety of 3-(2,4 dimethoxybenzylidene anabaseine) and related compounds.

The purpose of the trial is to lay the groundwork for Phase III investigation. If this trial finds that 3-(2,4 dimethoxybenzylidene anabaseine) has effects at a safe dose, without tachyphylaxis, then the investigators intend to proceed to a Phase III trial, where the clinical importance of this effect can be measured.

The trial will be a double blind trial with placebo control. The order of doses and placebo will be randomized.

The Phase 1 study was completed in January, 2005, with 12 non-smoking schizophrenics subjects. The subjects were concurrently treated with neuroleptics throughout the study. They received 3 treatments, each for 1 day, in a double-blind crossover design. The treatments were 3-(2,4 dimethoxybenzylidene anabaseine) (150 mg + 75 mg 2 hours later), 3-(2,4 dimethoxybenzylidene anabaseine)(75 mg + 37.5 mg 2 hours later), and placebo. A significant effect on neurocognition, as measured by the Repeatable Battery for Assessment of Neuropsychological Status, and on sensory gating, as measured by P50 auditory evoked potentials was observed. Subjects reported no significant symptoms. One subject's white blood cell count decreased from just above normal limits on placebo to just below normal levels on 3-(2,4 dimethoxybenzylidene anabaseine)(150 + 75 mg 2 hours later). He did not receive further exposure to drug and his white blood cell count returned to normal at the next testing, 2 days later.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* Currently treated with neuroleptic drugs

Exclusion Criteria:

* Treatment with clozapine;
* Head injury or neurological condition;
* Cardiovascular disease;
* Substance abuse or dependence, including nicotine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (1):
- VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tregellas JR, Tanabe J, Rojas DC, Shatti S, Olincy A, Johnson L, Martin LF, Soti F, Kem WR, Leonard S, Freedman R. Effects of an alpha 7-nicotinic agonist on default network activity in schizophrenia. Biol Psychiatry. 2011 Jan 1;69(1):7-11. doi: 10.1016/j.biopsych.2010.07.004. Epub 2010 Aug 21. PMID 20728875
- [Derived] Freedman R, Olincy A, Buchanan RW, Harris JG, Gold JM, Johnson L, Allensworth D, Guzman-Bonilla A, Clement B, Ball MP, Kutnick J, Pender V, Martin LF, Stevens KE, Wagner BD, Zerbe GO, Soti F, Kem WR. Initial phase 2 trial of a nicotinic agonist in schizophrenia. Am J Psychiatry. 2008 Aug;165(8):1040-7. doi: 10.1176/appi.ajp.2008.07071135. Epub 2008 Apr 1. PMID 18381905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-four subjects were screened. Two were excluded because of abnormal laboratory values and one was excluded for a recent hospitalization. Thirty-one subjects were enrolled at two sites: The University of Colorado, Denver/Denver VA Medical Center (25 subjects) and The Maryland Psychiatric Research Center 6 subjects.
Pre-assignment Details: Subjects were administered 1 week of placebo to assess their ability to comply with BID dosing prior to administration of drug or placebo. There was a 1 week washout period between arms.
Groups:
- Placebo, Then DMXB-A 75, Then DMXB-A 150: Placebo then 3-(2,4-dimethoxybenzylidene) anabaseine 75 mg then 3-(2,4-dimethoxybenzylidene) anabaseine 150 mg
- DMXB-A 75, Then DMXB-A 150, Then Placebo: 3-(2,4-dimethoxybenzylidene) anabaseine 75 mg,then 3-(2,4-dimethoxybenzylidene) anabaseine 150 mg, then placebo
- DMXB-A 150 mg, Then Placebo, Then DMXB-A 75: 3-(2,4-dimethoxybenzylidene) anabaseine 150 mg, then placebo, then 3-(2,4-dimethoxybenzylidene) anabaseine 75 mg
Period: Baseline
Arm/Group | Placebo, Then DMXB-A 75, Then DMXB-A 150 | DMXB-A 75, Then DMXB-A 150, Then Placebo | DMXB-A 150 mg, Then Placebo, Then DMXB-A 75
Started | 10 | 10 | 9
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 0
Period: First Intervention (4 Weeks)
Arm/Group | Placebo, Then DMXB-A 75, Then DMXB-A 150 | DMXB-A 75, Then DMXB-A 150, Then Placebo | DMXB-A 150 mg, Then Placebo, Then DMXB-A 75
Started | 10 | 10 | 9
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Placebo, Then DMXB-A 75, Then DMXB-A 150 | DMXB-A 75, Then DMXB-A 150, Then Placebo | DMXB-A 150 mg, Then Placebo, Then DMXB-A 75
Started | 10 | 10 | 9
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Placebo, Then DMXB-A 75, Then DMXB-A 150 | DMXB-A 75, Then DMXB-A 150, Then Placebo | DMXB-A 150 mg, Then Placebo, Then DMXB-A 75
Started | 10 | 10 | 9
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Placebo, Then DMXB-A 75, Then DMXB-A 150 | DMXB-A 75, Then DMXB-A 150, Then Placebo | DMXB-A 150 mg, Then Placebo, Then DMXB-A 75
Started | 10 | 10 | 9
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 0
Period: Third Intervention (4 Weeks)
Arm/Group | Placebo, Then DMXB-A 75, Then DMXB-A 150 | DMXB-A 75, Then DMXB-A 150, Then Placebo | DMXB-A 150 mg, Then Placebo, Then DMXB-A 75
Started | 10 | 10 | 9
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DMXB-A 75, Then DMXB- 150, Then Placebo: Overall number of baseline participants 10
  Age, continuous
- Placebo, Then DMXB-A 75, Then DMXB-A 150: Overall number of baseline participants 10
  Age , continuous
- DMXB-A 150, Then Placebo, Then DMXB-A 75: Overall number of baseline participants 9
  Age, continuous
- Total: Total of all reporting groups
Arm/Group | DMXB-A 75, Then DMXB- 150, Then Placebo | Placebo, Then DMXB-A 75, Then DMXB-A 150 | DMXB-A 150, Then Placebo, Then DMXB-A 75 | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (10.3) | 40.5 (9.8) | 43.2 (10.4) | 41.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 7 | 21
  Male | 3 | 3 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Neurocognitive Performance
Description: The measurement of neurocognitive performance on 6 domains, speed of processing, attention/vigilance, working memory, verbal learning, visual learning and reasoning/problem solving. Each domain is compared to a normative sample of schizophrenia subjects and the performance is determined and compared by a T-Test to the subjects baseline performance to determine the effect of drug or placebo. The scale is the National Institute of Mental Health Measurement and Treatment Research to Improve Cognition in Schizophrenia Neurocognitive Consensus Combined Battery, range 0-100. A higher score indicates better performance.
Time Frame: 1 month
Population: change from baseline in cognitive performance as measured by a t-test at 4 weeks after taking the drug or placebo
Measure: Mean (Standard Deviation); unit: t-score change from baseline
Groups:
- Placebo: Change in t-score from baseline performance on neurocognitive measures when taking placebo for 4 weeks
- 3-(2,4-dimethoxybenzylidene) Anabaseine 75 mg: Change in t-scores from baseline neurocognitive performance when taking 3-(2,4-dimethoxybenzylidene) anabaseine 75 mg p.o. BID for 4 weeks
- 3-(2,4-dimethoxybenzylidene) Anabaseine 150 mg: Change in t-scores from baseline neurocognitive performance when taking3-(2,4-dimethoxybenzylidene) anabaseine 150 mg p.o BID for 4 weeks
Arm/Group | Placebo | 3-(2,4-dimethoxybenzylidene) Anabaseine 75 mg | 3-(2,4-dimethoxybenzylidene) Anabaseine 150 mg
Number analyzed (Participants) | 29 | 29 | 29
t-score change from baseline | 4.5 (7.3) | 6.1 (9.4) | 7.6 (10.6)

2. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS)
Description: The Scale for the Assessment of Negative Symptoms measures the measure negative symptoms in schizophrenia by measuring the domains of anhedonia, alogia, avolition and anhedonia in schizophrenia on a scale from 1 to 20 that sums the global scores of all 4 domains, each of which are rated on a scale of 1-5. Higher scores indicate greater severity of negative symptoms
Time Frame: 1 month
Population: change in the total scale score from baseline measure with administration of either drug or placebo
Measure: Mean (Standard Deviation); unit: units on a scale change from baseline
Groups:
- 3-2,4 Dimethoxybenzylidene 75 mg: change in total scale for the assessment of negative symptoms at baseline after taking 3-2,4 dimethoxybenzylidene 75 mg BID for 4 weeks
- 3-2,4 Dimethoxybenzylidene 150 mg: change in total scale for the assessment of negative symptoms at baseline after taking 3-2,4 dimethoxybenzylidene BID 150 mg for 4 weeks
- Placebo: change in total scale for the assessment of negative symptoms at baseline after taking placebo BID for 4 weeks
Arm/Group | 3-2,4 Dimethoxybenzylidene 75 mg | 3-2,4 Dimethoxybenzylidene 150 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29
units on a scale change from baseline | 6.1 (9.4) | 7.6 (10.6) | 4.6 (6.5)

ADVERSE EVENTS:
Time Frame: Four weeks for each intervention
Description: Safety population included all participants who received at least one dose of intervention
Groups:
- DMXB-A 75 mg: 3-(2,4 dimethoxybenzylidene) 75 mg p.o. BID for 4 weeks
- DMXBA 150 mg: 3-(2,4 dimethoxybenzylidene) 150 mg p.o. BID for 4 weeks
- Placebo: Placebo p.o. BID for 4 weeks
Arm/Group | DMXB-A 75 mg | DMXBA 150 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 29/29 | 29/29 | 29/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DMXB-A 75 mg (N=29) | DMXBA 150 mg (N=29) | Placebo (N=29)
rash (Skin and subcutaneous tissue disorders) | 2/10 (2) | 3 (3) | 0 (0)
insomnia (Psychiatric disorders) | 5 (5) | 0 (0) | 2 (2)
sedation (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2)
malaise (General disorders) | 3 (3) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 0 (0) | 6 (6) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
restlessness (Nervous system disorders) | 3 (3) | 6 (6) | 2 (2)
nervousness (Psychiatric disorders) | 9 (9) | 5 (5) | 6 (6)
visual changes (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
tinnitus (Ear and labyrinth disorders) | 4 (4) | 0 (0) | 6 (6)
dry mouth (General disorders) | 3 (3) | 3 (3) | 2 (2)
drooling (General disorders) | 3 (3) | 4 (4) | 3 (3)
change in taste (General disorders) | 0 (0) | 2 (2) | 0 (0)
diaphoresis (General disorders) | 0 (0) | 0 (0) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 4 (4)
nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4)
diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (4)
flatulence (Gastrointestinal disorders) | 6 (6) | 4 (4) | 4 (4)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2)
constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4)
enuresis (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
limb pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 2 (2)
stiffness (Nervous system disorders) | 5 (5) | 3 (3) | 3 (3)
tremor (Nervous system disorders) | 6 (6) | 6 (6) | 5 (5)
parasthesias (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2)
hallucinations (Psychiatric disorders) | 9 (9) | 9 (9) | 8 (8)
delusions (Psychiatric disorders) | 9 (9) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes